CLINICAL TRIAL: NCT00920764
Title: A Phase 2a, Prospective, Randomized, Double-blind, Placebo-controlled Multicenter Study to Evaluate the Safety and Efficacy of Atrasentan on Reducing Albuminuria in Type 2 Diabetic Nephropathy Subjects Who Are Currently Being Treated With an Renin-Angiotensin System Inhibitor
Brief Title: A Study of Atrasentan on Reducing Albuminuria in Type 2 Diabetic Nephropathy Treated With Renin-Angiotensin System Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-815
Record Dates: First submitted 2009-06-11; First posted 2009-06-15 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2013-01

CONDITIONS: Chronic Kidney Disease; Diabetic Nephropathy
Keywords: CKD Stages 3&4; Endothelin antagonist; Proteinuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetic Nephropathies; Proteinuria | interventions — Atrasentan; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Active Comparator)
  Interventions: Drug: 1.75 mg Atrasentan QD
- B (Active Comparator)
  Interventions: Drug: 0.25 mg Atrasentan QD
- C (Active Comparator)
  Interventions: Drug: 0.75 mg Atrasentan QD
- D (Placebo Comparator)
  Interventions: Drug: Placebo for Atrasentan 0.2 mg/mL solution

INTERVENTIONS:
Drug: Placebo for Atrasentan 0.2 mg/mL solution — 10 mL oral solution, daily, 8 weeks
  Arms: D
Drug: 0.25 mg Atrasentan QD — 10 mL oral solution, daily, 8 weeks
  Arms: B
Drug: 0.75 mg Atrasentan QD — 10 mL oral solution, daily, 8 weeks
  Arms: C
Drug: 1.75 mg Atrasentan QD — 10 mL oral solution, daily, 8 weeks
  Arms: A

SUMMARY:
The study objective is to investigate the effects of three low doses of atrasentan on urinary albumin/creatinine ratio (UACR) levels in subjects with Type 2 diabetic nephropathy.

Patients with Type 2 diabetes with nephropathy must be receiving a renin-angiotensin system inhibitor, such as an Angiotensin converting enzyme inhibitor (ACEi) or an Angiotensin II Receptor Blocker (ARB) for participation in this study. ACEi and ARB treatment are the standard of care for the management of proteinuria in Chronic Kidney Disease (CKD) patients.

ELIGIBILITY:
Inclusion Criteria:

* 1.Subject is >= 18 years old.
* 2.Subject has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), after the nature of the study has been explained and the subject has had the opportunity to ask questions. The informed consent must be signed before any study-specific procedures are performed.
* 3.Subject has Type 2 diabetes and has been treated with at least one anti-hyperglycemic medication within the 12 months prior to the Screening Phase.
* 4.Subject has been receiving a stable dose (i.e., same type and regimen) of angiotensin-converting enzyme inhibitors (ACEi) and/or angiotensin receptor blocking agents (ARB) for at least 2 months prior to the Screening Phase.
* 5.If female, subject must be not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy). The reason for non-childbearing potential must be specified in the subject's eCRF.
* 6.If male, subject must be surgically sterile or if sexually active and of childbearing potential, the site must document the lack of desire for future procreation and subject must agree to use a condom and a second reliable barrier of contraception from the Screening Visit through two months following completion of their participation in the study.
* 7.For entry into the Treatment Phase the subject must satisfy the following criteria based on Screening laboratory values:

  * a.Estimated GFR > 20 mL/min/1.73 m2 by simplified MDRD formula
  * b.UACR between 100 and 3000 mg/g as determined at the initial Screening visit or by the mean of the 2 morning void urine specimens obtained prior to the second Screening visit.
  * c.Serum albumin > 3.0 g/dL.
  * d.HbA1c <= 10%.
  * e.Pro-BNP <= 500pg/mL.
  * f.Negative urine pregnancy test for female subjects.

Exclusion Criteria:

* 1.Subject has a history of significant peripheral edema (2 + or greater), or facial edema unrelated to trauma, or a history of myxedema in the 6 months prior to Screening.
* 2.Subject receiving loop diuretics > 30 mg BID of furosemide or > 0.5 mg BID of bumetanide or > 25 mg BID of ethacrynic acid.
* 3.Subject has a history of pulmonary edema.
* 4.Subject has a history of pulmonary hypertension, chronic obstructive pulmonary disease, emphysema, pulmonary fibrous disease, asthma or other lung disease that requires oxygen.
* 5.Subject has a documented history of heart failure, defined as New York Heart Association (NYHA) Class II, III or IV heart failure.
* 6.Subject has a body mass index (BMI) > 40.
* 7.Subject has elevated liver enzymes (ALT and/or AST) > 1.5 x the upper limit of normal (ULN).
* 8.Subject has a hemoglobin < 9.5 g/dL.
* 9.Subject has a history of an allergic reaction or significant sensitivity to atrasentan or its excipients.
* 10.Subject has a history of a chronic gastrointestinal disease, which in the Investigator's opinion may cause significant GI malabsorption.
* 11.Subject has a history of secondary hypertension (i.e., renal artery stenosis, primary aldosteronism or pheochromocytoma).
* 12.Subject has poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg and or diastolic blood pressure ≥ 90 mmHg) or hypotension (systolic blood pressure <= 90 mmHg).
* 13.Subject has significant comorbidities (e.g., advanced malignancy, advanced liver disease) with a life expectancy less than 1 year.
* 14.Subject is expected to receive an increased dose of current RAAS inhibitor (ACEi, ARB, renin or aldosterone inhibitor) during the course of the study. Conversions from one product to another (e.g., ACEi to ARB) must be at equivalent doses.
* 15.Subject has clinically significant coronary artery disease (CAD) within 3 months prior to the Screening Period, defined as one of the following:

  * Hospitalization for MI or unstable angina; or
  * New onset angina with positive functional study or coronary angiogram revealing stenosis; or
  * Coronary revascularization procedure.
* 16.Subject has a history of viral or bacterial infection within 4 weeks of Screening or HIV infection.
* 17.Subject has scheduled or planned surgery with general anesthesia within 12 weeks of Screening Visit.
* 18.Subject has a history of drug or alcohol abuse within 6 months prior to the Screening Visit.
* 19.Subject has evidence of poor compliance with diet or medication that may interfere, in the Investigator's opinion, with adherence to the protocol.
* 20.Subject has received any investigational drug within 30 days prior to study drug administration.
* 21.For any reason, subject is considered by the Investigator to be an unsuitable candidate to receive atrasentan oral solution or is put at risk by study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to each post-baseline observation on UACR over the course of treatment period versus standard of care | Week 8 visit or final assessment

SECONDARY OUTCOMES:
Proportion of subjects achieving at least a 25% reduction in final UACR levels from baseline | Week 8 visit or final assessment
Proportion of subjects achieving at least a 40% reduction in final UACR levels from baseline | Week 8 visit or final assessment
Change from baseline to the final value in UACR, estimated glomerular filtration rate (eGFR), Neutrophil Gelatinase-Associated Lipocalin (NGAL) | Week 8 visit or final assessment
Change from baseline to each weekly measurement in NGAL | Week 8 visit or final assessment

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Andress, Study Director — AbbVie
Locations (28):
- United States (24):
  - Site Reference ID/Investigator# 19386, Tempe, Arizona
  - Site Reference ID/Investigator# 25043, Azusa, California
  - Site Reference ID/Investigator# 23308, Los Angeles, California
  - Site Reference ID/Investigator# 25430, Los Angeles, California
  - Site Reference ID/Investigator# 20421, San Diego, California
  - Site Reference ID/Investigator# 22442, San Diego, California
  - Site Reference ID/Investigator# 21061, Whittier, California
  - Site Reference ID/Investigator# 16572, Yuba City, California
  - Site Reference ID/Investigator# 26142, Coral Gables, Florida
  - Site Reference ID/Investigator# 16567, Hudson, Florida
  - Site Reference ID/Investigator# 16577, Pembroke Pines, Florida
  - Site Reference ID/Investigator# 25242, Pembroke Pines, Florida
  - Site Reference ID/Investigator# 16569, Rockville, Maryland
  - Site Reference ID/Investigator# 16574, Omaha, Nebraska
  - Site Reference ID/Investigator# 20221, Buffalo, New York
  - Site Reference ID/Investigator# 16576, Greenville, North Carolina
  - Site Reference ID/Investigator# 16573, Morehead City, North Carolina
  - Site Reference ID/Investigator# 26143, Statesville, North Carolina
  - Site Reference ID/Investigator# 19383, Bethlehem, Pennsylvania
  - Site Reference ID/Investigator# 26365, Orangeburg, South Carolina
  - Site Reference ID/Investigator# 16571, San Antonio, Texas
  - Site Reference ID/Investigator# 16566, San Antonio, Texas
  - Site Reference ID/Investigator# 19384, San Antonio, Texas
  - Site Reference ID/Investigator# 24542, Fairfax, Virginia
- Puerto Rico (4):
  - Site Reference ID/Investigator# 16564, Las Piedras
  - Site Reference ID/Investigator# 19381, Ponce
  - Site Reference ID/Investigator# 16563, San Juan
  - Site Reference ID/Investigator# 16562, San Juan

REFERENCES:
- [Background] Perez-Gomez MV, Sanchez-Nino MD, Sanz AB, Martin-Cleary C, Ruiz-Ortega M, Egido J, Navarro-Gonzalez JF, Ortiz A, Fernandez-Fernandez B. Horizon 2020 in Diabetic Kidney Disease: The Clinical Trial Pipeline for Add-On Therapies on Top of Renin Angiotensin System Blockade. J Clin Med. 2015 Jun 18;4(6):1325-47. doi: 10.3390/jcm4061325. PMID 26239562